CLINICAL TRIAL: NCT04816513
Title: An Open-label, Randomized, Parallel-group Study to Assess the Bioequivalence of Ustekinumab Following a Single Subcutaneous Administration by Two Different Injection Devices in Healthy Participants
Brief Title: A Study to Assess the Bioequivalence of Ustekinumab by Two Different Injection Devices in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108948; CNTO1275EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ustekinumab (Using Reference Device) (Active Comparator): Participants will receive a single subcutaneous (SC) injection of ustekinumab in Device 1 as a reference device on Day 1.
  Interventions: Drug: Ustekinumab
- Ustekinumab (Using Test Device) (Experimental): Participants will receive a single SC injection of ustekinumab in Device 2 as a test device on Day 1.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab will be administered as SC injection.
  Other Names: CNTO1275, STELARA

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) and bioequivalence (BE) of ustekinumab administered by a single subcutaneous (SC) injection with Device 1 or Device 2 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be a non-user or a light user of tobacco products (not smoke more than 10 cigarettes or equivalent a day for at least 6 months prior to screening), including all nicotine use, example, cigarettes (including e-cigarettes or the equivalent of e-cigarettes), cigars, chewing tobacco, patch, gum
* Body weight within the range of 50.0 kilograms (kg) to 90.0 kg, inclusive and body mass index within the range of 18 kilograms per meter square (kg/m^2) to 30 kg/m^2 (inclusive)
* A female participant must have a negative pregnancy test result at screening and baseline (Day -1) and while enrolled in this study
* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 12 weeks after study intervention
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 12 weeks after receiving the last dose of study intervention

Exclusion Criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurologic or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* History of malignancy before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Has previously received ustekinumab
* Received an investigational intervention (including investigational vaccines or devices) or used an invasive investigational device within 30 days or 5 half lives before screening or is currently enrolled in an investigational study
* Has a current chronic infection, prior history of recurrent infection, or an active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentrations (Cmax) of Ustekinumab | Up to Day 85
  Cmax is maximum observed serum concentration of ustekinumab.
Area Under the Serum Concentration Versus Time Curve from Time Zero to Infinity (AUC [0-Infinite]) | Up to Day 85
  AUC (0-Infinite) defined as area under the serum concentration versus time curve from time zero to infinity with extrapolation of the terminal phase will be evaluated.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 85
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with AEs Related to the Injection or at the Injection Site | Up to Day 85
  Number of participants with AEs related to injection or at the injection site will be reported. Symptoms such as erythema, induration and pruritis that in the opinion of the investigator may be associated with the administration, will be captured as an AE (example, injection-site erythema, injection-site induration, injection-site pruritis or injection-site pain.
Number of Participants with Abnormalities in Vital Signs | Up to Day 85
  Number of participants with abnormalities in vital signs (temperature [oral], pulse/heart rate, respiratory rate, and blood pressure [systolic and diastolic]) will be reported.
Number of Participants with Abnormalities in Physical Examinations (PE) | Up to Day 85 (for full PE) and up to Day 57 (for brief PE)
  Number of participants with abnormalities in physical examinations (full and brief) will be reported. Full physical examinations will include a review of the following body systems: general appearance; thorough skin and oral mucosa evaluation; eyes, ears, nose, and throat; cardiovascular; respiratory; abdomen; peripheral pulsation; lymph nodes; neurologic (including examination for muscle strength and sensory exam); musculoskeletal; head, neck, and thyroid. A brief physical examination includes basic assessment of general appearance, respiratory and cardiovascular systems and the assessment of the skin at the administration area.
Number of Participants with Abnormalities in Laboratory Tests | Up to Day 85
  Number of participants with abnormalities in laboratory tests (serum chemistry and hematology and urinalysis) will be reported.
Number of Participants with Antibodies to Ustekinumab | Up to Day 85
  Number of participants with antibodies to ustekinumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Celerion, Tempe, Arizona
  - Celerion, Lincoln, Nebraska
  - PRA Health Sciences, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency